CLINICAL TRIAL: NCT03886142
Title: Efficacy of Genicular Nerve Radiofrequency Ablation Versus Intra-Articular Platelet Rich Plasma in Chronic Knee Osteoarthritis; a Randomized Clinical Trial
Brief Title: Platelet Rich Plasma Versus Radio Frequency for Chronic Knee Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009923
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteo Arthritis Knee; Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: patients with chronic knee osteoarthritis non res ponders to conventional medical treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency (Active Comparator): genicular nerves pulsed radiofrequency
  Interventions: Procedure: radiofrequency
- intra-articular platelet rich plasma (Active Comparator): injection of platelet rich plasma in the affected joint
  Interventions: Procedure: platelet rich plasma injection

INTERVENTIONS:
Procedure: radiofrequency — radiofrequency of the genicular nerves
  Arms: radiofrequency
Procedure: platelet rich plasma injection — intra articular injection of platelet rich plasma
  Arms: intra-articular platelet rich plasma

SUMMARY:
Osteoarthritis (OA) affects aged above 45 years. RF has been used for several painful conditions. There have been a few attempts to use RF current for the treatment of painful conditions of joints of the extremities. It was also used for the treatment of painful conditions of the hip joint.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis knee

Exclusion Criteria:

* coaguloapthy
* patient refusal

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
pain visual analog scale | 12 months
  assessment of visual analog scale (VAS) VAS of zero means no pain, and 10 means sever pain

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt